CLINICAL TRIAL: NCT03018340
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of Adjunctive Pimavanserin in Major Depressive Disorder
Brief Title: Study to Evaluate the Efficacy and Safety of Adjunctive Pimavanserin in Major Depressive Disorder (CLARITY)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-042
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Adjunctive Treatment of Major Depressive Disorder
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pimavanserin 34 mg + SSRI/SNRI (Experimental): Drug- pimavanserin, 34 mg, taken as two 17 mg tablets, once daily by mouth All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
  Interventions: Drug: Pimavanserin
- Placebo + SSRI/SNRI (Placebo Comparator): Placebo, taken as two tablets, once daily by mouth All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg, tablet, taken as two 17 mg tablets, once daily by mouth All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
  Arms: Pimavanserin 34 mg + SSRI/SNRI
Other: Placebo — Placebo, taken as two tablets, once daily by mouth All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
  Arms: Placebo + SSRI/SNRI

SUMMARY:
To assess the efficacy of pimavanserin compared to placebo when given adjunctively to a selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant as treatment of patients with Major Depressive Disorder (MDD) and an inadequate response to antidepressant therapy

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged 18 years and above
2. A clinical diagnosis of major depressive disorder (MDD)
3. Is being treated with one of the following SSRI or SNRI antidepressants as monotherapy:

   * Citalopram
   * Escitalopram
   * Paroxetine
   * Fluoxetine
   * Sertraline
   * Duloxetine
   * Venlafaxine
   * Desvenlafaxine
   * Venlafaxine XR
4. Has a history of inadequate response to antidepressant treatments

Exclusion Criteria:

1. Patient has a psychotic disorder other than MDD
2. Patient has current evidence of a serious and/or unstable neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the program
3. Patient has a history or symptoms of long QT syndrome

Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - UAB, Birmingham, Alabama
  - Woodland Research Northwest, Rogers, Arkansas
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy San Diego, National City, California
  - Pacific Research Partners, LLC, Oakland, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Meridien Research, Bradenton, Florida
  - CNS Health care (Jacksonville), Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - CNS Health care (Orlando), Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Alam Medical Research, INC, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - KUMC, Wichita, Kansas
  - St. Louis Clinical Trials, St Louis, Missouri
  - Altea Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Portland, Oregon
  - UPenn, Philadelphia, Pennsylvania
  - BTC of Lincoln, Lincoln, Rhode Island
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - UTSW, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Ericksen Research & Development, Clinton, Utah
  - IPC Research, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jha MK, Fava M, Freeman MP, Thase ME, Papakostas GI, Shelton RC, Trivedi MH, Dirks B, Liu K, Stankovic S. Effect of Adjunctive Pimavanserin on Sleep/Wakefulness in Patients With Major Depressive Disorder: Secondary Analysis From CLARITY. J Clin Psychiatry. 2020 Dec 1;82(1):20m13425. doi: 10.4088/JCP.20m13425. PMID 33264819
- [Derived] Fava M, Dirks B, Freeman MP, Papakostas GI, Shelton RC, Thase ME, Trivedi MH, Liu K, Stankovic S. A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of Adjunctive Pimavanserin in Patients With Major Depressive Disorder and an Inadequate Response to Therapy (CLARITY). J Clin Psychiatry. 2019 Sep 24;80(6):19m12928. doi: 10.4088/JCP.19m12928. PMID 31556975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Stage 1, pts were randomized to pimavanserin or placebo (1:3). At the end of Stage 1, placebo pts not responding to treatment were rerandomized (1:1) in Stage 2; all other pts continued in Stage 2 the initial randomized treatment.
Groups:
- Pimavanserin 34 mg + SSRI/SNRI: Patients randomized to Pimavanserin at the beginning of Stage 1. Patients on Pimavanserin remained on their assigned treatment throughout Stage 1 and 2 of the study.
  Pimavanserin 34 mg (2 x 17 mg), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
- Placebo + SSRI/SNRI: Patients randomized to Placebo at the beginning of Stage 1. This group includes all patients randomized to placebo in Stage 1, irrespective of response in Stage 1 and later rerandomization to Pimavanserin or Placebo in Stage 2.
  Placebo (2 x Placebo tablets), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
Period: Overall Study
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI | Placebo + SSRI/SNRI
Started | 52 | 155
Completed | 44 | 125
Not Completed | 8 | 30
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-compliance with study drug/procedure | 3 | 4
Not completed — Lost to Follow-up | 1 | 7
Not completed — Protocol Violation | 3 | 7
Not completed — Not further specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients randomized. Baseline measures are shown for Stage 1 baseline, as Stage 2 baseline included the subset of Stage 1 patients meeting re-randomization criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI | Placebo + SSRI/SNRI | Total
Number analyzed (Participants) | 52 | 155 | 207
Age, Customized [Count of Participants; unit: Participants]
  18-40 years | 14 | 55 | 69
  >40 years | 38 | 100 | 138
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 108 | 151
  Male | 9 | 47 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 7 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 31 | 40
  White | 38 | 111 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 5 in the HAMD-17 Total Score
Description: The Hamilton Rating Scale for Depression (HAMD-17) is a 17-item scale to assess depression. The HAMD-17 consists of 8 items with a score on a 3 point scale and 9 items with a score on a 5 point scale. Each item is rated from least (0) to most frequent or most severe, as applicable, with highest scores of 2 to 4, depending on the item. Items are summed up to calculate the HAMD-17 total score. The total score ranges from 0 to 52. A higher total score indicates more severe depression.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: FAS Stage 1: pts randomized to Stage 1, received ≥1 dose of study drug in Stage 1, and had a baseline value and ≥1 post-baseline value for HAMD-17 total score in Stage 1.
  FAS Stage 2: pts randomized to Stage 2, received ≥1 dose of study drug in Stage 2, and had a baseline value and ≥1 post-baseline value for HAMD-17 total score in Stage 2.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Pimavanserin 34 mg + SSRI/SNRI, Stage 1: Patients randomized to Pimavanserin at the beginning of Stage 1. Patients on Pimavanserin remained on their assigned treatment throughout Stage 1 and 2 of the study. Pimavanserin 34 mg (2 x 17 mg), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
- Placebo + SSRI/SNRI, Stage 1: Patients randomized to Placebo at the beginning of Stage 1. This group includes all patients randomized to placebo in Stage 1, irrespective of response in Stage 1 and later rerandomization to Pimavanserin or Placebo in Stage 2. Placebo (2 x Placebo tablets), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
- Pimavanserin 34 mg + SSRI/SNRI, Stage 2: Patients rerandomized to Pimavanserin 34 mg at the beginning of Stage 2. Patients represent a subset of the placebo patients not responding to treatment (by protocol-defined criteria) in Stage 1, who were then randomly assigned (1:1) to pimavanserin or placebo in Stage 2. Pimavanserin 34 mg (2 x 17 mg tablets), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
- Placebo + SSRI/SNRI, Stage 2: Patients rerandomized to Placebo at the beginning of Stage 2. Patients represent a subset of the placebo patients not responding to treatment (by protocol-defined criteria) in Stage 1 who were then randomly assigned (1:1) to pimavanserin or placebo in Stage 2. Placebo (2 x placebo tablets), once daily by mouth. All patients continued to receive selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) antidepressants at a stable dose for the duration of the study.
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 22.9 (0.62) | 22.0 (0.34) | 20.3 (0.83) | 20.4 (0.79)
  Change from BL to Week 5: number analyzed (Participants) | 45 | 127 | 29 | 24
  Change from BL to Week 5 | -11.9 (1.14) | -7.1 (0.55) | -2.8 (0.75) | -3.2 (1.17)
Statistical Analysis 1: Comparison: Pimavanserin 34 mg + SSRI/SNRI, Stage 1 vs Placebo + SSRI/SNRI, Stage 1 vs Pimavanserin 34 mg + SSRI/SNRI, Stage 2 vs Placebo + SSRI/SNRI, Stage 2; This is the primary statistical comparison for Stage 1 and Stage 2 combined; Test type: Superiority; p = 0.0390, Mixed Models Analysis; Difference in weighted MMRM LSMs = -1.7, 95% CI 2-sided [-3.4 to -0.1], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Pimavanserin 34 mg + SSRI/SNRI, Stage 1 vs Placebo + SSRI/SNRI, Stage 1; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Difference in MMRM LSMs = -4.0, 95% CI 2-sided [-6.1 to -1.9], Standard Error of Mean 1.09
Statistical Analysis 3: Comparison: Pimavanserin 34 mg + SSRI/SNRI, Stage 2 vs Placebo + SSRI/SNRI, Stage 2; Test type: Superiority; p = 0.6940, Mixed Models Analysis; Difference in MMRM LSMs = 0.5, 95% CI 2-sided [-2.1 to 3.1], Standard Error of Mean 1.30

2. Secondary Outcome: Change From Baseline to Week 5 in the SDS Total Score
Description: The Sheehan Disability Scale is a 3-item patient-facing questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point scale from 0 (no impairment) to 10 (most severe). The total SDS score ranges from 0 to 10. It is calculated as the arithmetic mean of the scores for all 3 items. A higher score indicates greater disability.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: Stage 1: pts randomized to Stage 1, received ≥1 dose of study drug in Stage 1, and had a baseline value and ≥1 post-baseline value for HAMD-17 total score in Stage 1.
  Stage 2: pts randomized to Stage 2, received ≥1 dose of study drug in Stage 2, and had a baseline value and ≥1 post-baseline value for HAMD-17 total score in Stage 2.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Basline (BL) | 6.365 (0.2996) | 6.519 (0.1716) | 5.753 (0.3314) | 5.747 (0.4191)
  Change from BL to Week 5: number analyzed (Participants) | 45 | 127 | 29 | 24
  Change from BL to Week 5 | -3.229 (0.4436) | -2.026 (0.2233) | -0.890 (0.2798) | -0.507 (0.3288)

3. Secondary Outcome: Treatment Response and Remission Rates at the End of 5-week Treatment Period
Description: The Hamilton Rating Scale for Depression (HAMD-17) is a 17-item scale to assess depression. Each item is rated from least (0) to most frequent or most severe, as applicable, with highest scores of 2 to 4 depending on the item. Items are summed up to calculate the HAMD-17 total score. A higher total score indicates more severe depression.
  Treatment response was defined as a reduction from Baseline in HAMD-17 total score of >=50%.
  Remission was defined as a HAMD-17 total score <=7.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
Participants
  Treatment responders Week 5 | 27 | 38 | 2 | 2
  Remission rate Week 5 | 12 | 17 | 1 | 1

4. Secondary Outcome: Change From Baseline to Week 5 in CGI-S Total Score
Description: The Clinical Global Impression-Severity Scale is a 1-item scale, used to rate the severity of the disorder from 0 (not assessed) to 7 (among the most extremely ill patients). A higher CGI-I score denotes more severe depression.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 4.6 (0.09) | 4.4 (0.05) | 4.1 (0.16) | 4.1 (0.14)
  Change from BL to Week 5: number analyzed (Participants) | 44 | 127 | 29 | 24
  Change from BL to Week 5 | -2.0 (0.21) | -1.1 (0.10) | -0.5 (0.13) | -0.5 (0.23)

5. Secondary Outcome: CGI-I Score at Week 5
Description: The Clinical Global Impression- Improvement scale is a 1-item scale, used to rate the global improvement of the patient since beginning of the study from 0 (not assessed) to 7 (very much worse). A higher CGI-I score denotes less improvement in depression.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 44 | 127 | 29 | 24
score on a scale | 2.2 (0.17) | 2.8 (0.10) | 3.0 (0.18) | 3.1 (0.19)

6. Secondary Outcome: Change From Baseline to Week 5 in SF-12 Score
Description: The 12-Item Short Form Health Survey is a patient-reported outcome measure that addresses 8 domains of physical functioning, role - physical, bodily pain, general health perceptions, vitality, social functioning, role - emotional, and mental health. Composite scores were obtained representing physical health and mental health composite summaries, Physical Component Summary (PCS) and Mental Component Summary (MCS), respectively. An algorithm was used to generate PCS and MCS for comparison to normative data. In normative data, the mean score was set to 50; thus, scores >50 indicate better physical or mental health than the mean and scores <50 indicate worse health. A higher score is indicative of a better health state.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 151 | 29 | 29
score on a scale
  PCS baseline (BL) | 49.587 (1.7918) | 48.783 (0.9845) | 46.945 (2.0961) | 48.994 (2.0596)
  PCS change from BL to Week 5 | -0.981 (1.1036) | -0.726 (0.7095) | -0.546 (1.4718) | 1.811 (1.2081)
  MCS baseline (BL) | 23.113 (1.2848) | 24.004 (0.6570) | 27.557 (1.4023) | 28.524 (1.5909)
  MCS change from BL to Week 5 | 16.146 (1.9531) | 7.989 (0.8137) | 3.566 (1.5421) | 0.578 (1.4600)

7. Secondary Outcome: Change From Baseline to Week 5 in DAI-10 Score
Description: The Drug Attitude Inventory-10 is a 6-item patient-facing questionnaire to evaluate a patient's perceptions and experiences of treatment. It contains 6 items that a patient who is fully adherent to prescribed medication would answer as "True," and 4 items that a patient who is fully adherent would rate as "False." Scores are allocated to each answer and the total score is calculated as the sum. A correct answer is scored +1 and an incorrect answer is scored -1. The total score ranges from -10 to 10 and is the sum of pluses and minuses. A positive total score indicates a positive subjective response (adherent) and a negative total score indicates a negative subjective response (nonadherent). Higher scores denoted better adherence.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 4.2 (0.61) | 4.4 (0.34) | 5.1 (0.68) | 4.8 (0.70)
  Change from BL to Week 5 | 1.4 (0.56) | 0.5 (0.26) | 0.6 (0.66) | 0.3 (0.50)

8. Secondary Outcome: Change From Baseline to Week 5 in KSS Score
Description: The Karolinska Sleepiness Scale is a patient-facing 1-item scale that measures the patient's drowsiness. Scoring is based on a 9-point verbally anchored scale ranging from "extremely alert" (1) to "very sleepy, great effort to keep awake, fighting sleep" (9). Higher scores denote more drowsiness.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 6.7 (0.19) | 6.6 (0.14) | 6.7 (0.29) | 6.1 (0.30)
  Change from BL to Week 5: number analyzed (Participants) | 45 | 127 | 29 | 24
  Change from BL to Week 5 | -1.9 (0.33) | -0.4 (0.18) | -0.5 (0.29) | -0.2 (0.29)

9. Secondary Outcome: Change From Baseline to Week 5 in MGH-SFI Score
Description: The Massachusetts General Hospital Sexual Functioning Index is a patient-facing questionnaire that quantifies sexual dysfunction into 5 functional domains ("interest in sex," "sexual arousal," "ability to achieve orgasm," "ability to maintain erection" [males only], and "sexual satisfaction"). Patients rate each item using a 6-point scale ranging from 1 (good function) to 6 (poor function). The MGH-SFI score is calculated as the arithmetic mean of the item scores for the 5 domains. The mean MGH-SFI score ranges from a minimum value of 1 to a maximum value of 6. Higher scores denotes worse sexual dysfunction.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 4.642 (0.1967) | 4.457 (0.1176) | 4.678 (0.2269) | 4.264 (0.2893)
  Change from BL to Week 5 | -0.830 (0.1814) | -0.155 (0.0807) | -0.472 (0.1580) | -0.183 (0.1085)

10. Secondary Outcome: Change From Baseline to Week 5 in BIS-11 Score
Description: The Barratt Impulsiveness Scale-11 is a questionnaire for assessment of the personality/behavioral construct of impulsiveness. It is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Items are scored on a 4-point scale from Rarely/Never (1) to Almost Always/Always (4). Items are summed up to calculate the total score. The BIS-11 total score ranges from 30 to 120. Higher scores denotes more impulsiveness.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 72.5 (1.53) | 70.0 (0.92) | 65.9 (1.79) | 70.3 (1.86)
  Change from BL to Week 5: number analyzed (Participants) | 45 | 126 | 28 | 24
  Change from BL to Week 5 | -4.2 (1.10) | -2.8 (0.72) | -1.4 (0.87) | 1.7 (1.33)

11. Secondary Outcome: Change From Baseline to Week 5 in SIS Score
Description: The Sheehan Irritability Scale is a 7-item patient-reported outcome measure to measure the frequency, severity, and impairment associated with irritability in psychiatric patients. It includes items on: irritability, frustration, edginess/ impatience/ overreaction, moodiness, anger with self, anger with others, and temper. Items are answered on an 11-point rating scale where higher scores indicated greater severity (0=not at all, 10=extremely). Item responses are summed into a total score (range=0-70). Higher scores mean higher irritability.
Time Frame: Baseline, 5 weeks and 10 weeks during Stage 1 and Stage 2, respectively
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
Number analyzed (Participants) | 51 | 152 | 29 | 29
score on a scale
  Baseline (BL) | 38.9 (2.04) | 38.8 (1.22) | 35.2 (2.45) | 36.6 (3.19)
  Change from BL to Week 5: number analyzed (Participants) | 45 | 126 | 28 | 24
  Change from BL to Week 5 | -19.4 (2.97) | -10.8 (1.42) | -4.8 (2.06) | -6.6 (2.77)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Safety analysis set Stage 1: all pts randomized to Stage 1 and received ≥1 dose of study drug in Stage 1 Safety analysis set Stage 2: all pts randomized to Stage 2 and received ≥1 dose of study drug in Stage 2
  AEs were summarized for the Safety analysis set Stage 1 (5 weeks) and for the Safety analysis set Stage 2 (5 weeks) separately.
  Patients in Stage 1 and 2 do not add up, as patients in Stage 2 are a subset of placebo non-responders from Stage 1.
Arm/Group | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 | Placebo + SSRI/SNRI, Stage 1 | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 | Placebo + SSRI/SNRI, Stage 2
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/155 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/155 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 22/52 | 36/155 | 6/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 (N=52) | Placebo + SSRI/SNRI, Stage 1 (N=155) | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 (N=29) | Placebo + SSRI/SNRI, Stage 2 (N=29)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin 34 mg + SSRI/SNRI, Stage 1 (N=52) | Placebo + SSRI/SNRI, Stage 1 (N=155) | Pimavanserin 34 mg + SSRI/SNRI, Stage 2 (N=29) | Placebo + SSRI/SNRI, Stage 2 (N=29)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 7 (8) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 14 (15) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 9 (9) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Interpretation of Stage 2 results is limited by the reduced number of patients vs initial projections anticipated by the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03018340/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03018340/SAP_001.pdf